CLINICAL TRIAL: NCT02849106
Title: Predictive Response to Chemotherapy (FOLFOX or FOLFIRI) by ex Vivo Culture 3D Technique in Metastatic Colorectal Cancer: a Preliminary Study
Brief Title: Predictive Response to Chemotherapy (FOLFOX or FOLFIRI) by ex Vivo Culture 3D Technique in Metastatic Colorectal Cancer
Acronym: CULTURE3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2009-08
Record Dates: First submitted 2016-07-13; First posted 2016-07-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
Keywords: 3D culture; chemogram; FOLFOX; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biopsy to obtain a chemogram (Experimental)
  Interventions: Procedure: biopsy to obtain a chemogram

INTERVENTIONS:
Procedure: biopsy to obtain a chemogram — All patients enrolled will have biopsies (on primary tumor or on a metastasis) before treatment in order to obtain a chemogram by ex vivo 3D culture cells

SUMMARY:
Prospective, open labelled, multicenter trial to evaluate the feasibility of ex vivo culture 3D (chemogram obtaining) on biopsies in order to estimate the predictive value of this technique for treatment response in patients treated by two different chemotherapies (FOLFOX or FOLFIRI) for colorectal cancer.

DETAILED DESCRIPTION:
The CULTURE 3D study is a prospective, open labelled, multicenter trial. The aim is to evaluate the feasibility of ex vivo culture 3D (chemogram) on biopsies in order to estimate the predictive value of this technique for treatment response in patients treated by two different chemotherapies (FOLFOX or FOLFIRI) for colorectal cancer.

Patients will have biopsies in a metastasis or in the primitive tumor before treatment. The sample will be used for a 3D ex vivo cells culture. A chemogram will be made based on cells proliferation data (Ki67) and apoptosis (M30).

Results from this chemogram will not interfere with the treatment combination choice.

The treatment response will be evaluated by the RECIST assessment and will be then compared to the chemogram.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or more
2. Colorectal cancer with synchronous or metachronous metastases
3. Metastasis and/or primitive tumor (in case of synchronous metastases) accessible to biopsy
4. Measurable metastatic disease (echography, CT and/or MRI, PET-FDG)
5. Indication for treatment with a combination including FOLFOX/FOLFIRI associated to an anti VEGF drug (Avastin)
6. No adjuvant chemotherapy for the primitive colorectal cancer and no line of chemotherapy for metastatic disease during the year prior to inclusion.
7. Life expectancy > 3 months (ECOG 0-1-2).
8. Informed and signed consent by the patient.

Exclusion Criteria:

1. Elevation of Carcinoembryonic antigen (CEA) without measurable metastatic disease
2. Medical contraindication to chemotherapy or biotherapy as FOLFOX/FOLFIRI or Avastin.
3. Treatment with FOLFOX/FOLFIRI and biotherapy anti-EGFR (epidermal growth factor receptor)(Erbitux) planned
4. Patient already enrolled in an other clinical trial with another first line of chemotherapy.
5. Pregnant women, breastfeeding or of childbearing age not taking contraceptive
6. Persons deprived of liberty.
7. Subject unable to make follow up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of interpretable chemogram | through study completion, an average of 1 year
  In ex vivo 3D culture from tumor biopsies, number of interpretable chemogram.

SECONDARY OUTCOMES:
Correlation between chemogram results obtained by 3D culture and RECIST 1.1 response assessement. | through study completion, an average of 1 year
  Number of chemogram showing the same response to treatment than patient RECIST 1.1 measured response.
Chemosensitivity evaluated on 3D culture. | through study completion, an average of 1 year
  on untreated and treated fragments : proliferating index (ki67) and apoptosis (M30) will be assessed.
time to obtain chemogram | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Mariani, MD, Principal Investigator — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Hôpital Lariboisière, Paris

IPD SHARING:
Plan to Share IPD: No